CLINICAL TRIAL: NCT02686034
Title: A Prospective, Multi-centre, Randomized, Double-blind, Sham-controlled Study of gammaCore® Non-invasive Vagus Nerve Stimulator (nVNS), for the Acute Treatment of Migraine
Brief Title: RCT of Non-Invasive Vagus Nerve Stimulation (nVNS) With gammaCore®, for the Acute Treatment of Migraine Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GM-16
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Migraine
Keywords: Migraine; Non-invasive vagus nerve stimulation; Vagus nerve stimulation; Vagal nerve stimulation; gammaCore; episodic migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gammaCore-S (Active Comparator): Treatment of up to 5 migraine attacks with the Active gammaCore-S non-invasive vagus nerve stimulator device which delivers a mild electrical signal in the vicinity of the vagus nerve
  Interventions: Device: gammaCore-S
- gammaCore-S Sham (Sham Comparator): Treatment of up to 5 migraine attacks with the Sham gammaCore-S non-invasive vagus nerve stimulator device which delivers a mild electrical signal in the vicinity of the vagus nerve
  Interventions: Device: gammaCore-S Sham

INTERVENTIONS:
Device: gammaCore-S — At onset of migraine pain, the subject self-administers a bilateral treatment with the gammaCore nVNS device (2 minutes on the right side, and 2 minutes on the left side). If their headache pain has not improved after 15 minutes, they administer another bilateral treatment. If they are not pain-free at 2 hours, they have the option to administer a third bilateral treatment, or take their usual rescue medication.
  Other Names: nVNS
  Arms: gammaCore-S
Device: gammaCore-S Sham — At onset of migraine pain, the subject self-administers a bilateral treatment with the gammaCore nVNS Sham device (2 minutes on the right side, and 2 minutes on the left side). If their headache pain has not improved after 15 minutes, they administer another bilateral treatment with the Sham device. If they are not pain-free at 2 hours, they have the option to administer a third bilateral treatment with the Sham device, or take their usual rescue medication.
  Other Names: sham nVNS
  Arms: gammaCore-S Sham

SUMMARY:
This study is a prospective, multi-centre, randomised, double-blind, sham-controlled investigation designed for comparison of two parallel treatment groups: gammaCore (active nVNS treatment) and a Sham device (control treatment), for the acute treatment of migraine attacks

DETAILED DESCRIPTION:
Period 1: 4-week observational run-in period; no stimulation treatment. Subjects use standard of care (SoC) medication to treat their migraine attacks, according to their individual prescriptions.

Period 2: 4-week randomized/controlled period. After the run-in period, subjects are randomized (1:1) to receive either an nVNS device or a sham device to treat up to 5 migraine attacks.

Period 3: 4-week open-label (active treatment) period. After the randomized period, subjects continue to the open-label period where all subjects receive an active gammaCore device to treat up to 5 migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18-75 years old.
2. Has been previously diagnosed with migraine (with or without aura) in accordance with the ICHD-3 Beta classification criteria.
3. Age of onset of migraines < 50 years old.
4. Experiences between 3-8 migraine attacks per month of moderate or severe intensity, and less than 15 headache days per month over the last 6 months.
5. Is able to distinguish migraine headaches from other headaches (e.g. tension type headache).
6. Agrees to withhold usual acute migraine medications until 2 hours after stimulation treatment with the study device.
7. Agrees not to initiate new or change existing migraine prophylaxis medication for the duration of the study, or receive nerve blocks or injections.
8. Agrees not to initiate new or change existing prophylactic medication for indications other than migraine that in the opinion of the Investigator may interfere with the study objectives (e.g. antidepressant, anti-convulsant, beta blockers, etc).
9. Has internet/web access for web-based e-Diary completion.
10. Agrees to use the study device as intended, comply with all study requirements including treatment, follow-up visits, record required study data in the subject diary, and complete study self-assessment questionnaires.
11. Is able to provide written informed consent.

Exclusion Criteria:

1. Experiences ≥ 15 headache days per month, including migraine, tension type headache, medication overuse headache, and other types of headache as defined in the ICHD-3 Beta classification.
2. Has a known history or suspicion of secondary headache.
3. Has previous diagnosis of medication overuse headache (MoH), which has reverted to episodic migraine within the last 6 months.
4. Has had surgical intervention for migraine prevention.
5. Has had a cervical vagotomy.
6. Has a structural abnormality (e.g. lymphadenopathy, neoplasm, previous surgery or abnormal anatomy), or pain (e.g. dysesthesia, neuralgia and/or cervicalgia) at the stimulation treatment site.
7. Has other significant pain problem (e.g. cancer pain, fibromyalgia or other head or facial disorder) that in the opinion of the Investigator may confound the study assessments.
8. Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, cochlear implant, sphenopalatine ganglion stimulator, or occipital nerve stimulator).
9. Has been implanted with metal cervical spine hardware or has a metallic implant near the stimulation treatment site.
10. Has failed an adequate trial (two months or greater) of at least 3 classes of a drug therapy for acute treatment of migraine.
11. Has initiated new, or changed existing medications for migraine prophylaxis in the previous 2 months.
12. Is using marijuana (including medical marijuana) for any indications, more than twice a month.
13. Currently takes simple analgesics or non-steroidal anti-inflammatory drugs (NSAIDS) greater than 15 days per month, or triptans, ergots or combined analgesics greater than 10 days per month.
14. Currently takes opioids greater than 2 days per month for headache relief or body pain.
15. Has undergone nerve block (occipital or other) in the head or neck within the last 2 months, or Botox injections within the last 6 months.
16. Has a concomitant medical condition that will require oral or injectable steroids during the study.
17. Has a history of intracranial aneurysm, intracranial haemorrhage, brain tumour or significant head trauma.
18. Has known or suspected severe cardiac disease (e.g. symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure(CHF), cerebrovascular disease (e.g. prior stroke or transient ischemic attack symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery), or uncontrolled high blood pressure (systolic >160, diastolic >100 after 3 repeated measurements within 24 hours).
19. Has a history of syncope or seizure (within the last 5 years).
20. Has a known history or suspicion of substance abuse or addiction (within the last 5 years).
21. Has psychiatric or cognitive disorder and/or behavioural problems which in the opinion of the clinician may interfere with the study.
22. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised (e.g. homeless, developmentally disabled, prisoner).
23. Is pregnant or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use an accepted form of birth control.
24. Is a relative or employee of the Investigator or the clinical study site.
25. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
26. Has previously used the gammaCore device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, PhD, Study Chair — IRCSS "National Neurological Institute C. Mondino" Foundation
Locations (10):
- Italy (10):
  - University Aldo Moro, Ospedale Pediatrico, Bari
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Ospedale Bellaria, Bologna
  - University Hospital of Careggi, Florence
  - Fondazione IRCCS Istituto Neurologico C. Besta, Milan
  - IRCSS "National Neurological Institute C. Mondino" Foundation, Pavia
  - S. Maria della Misericordia Hospital, Perugia
  - INM Neuromed IRCCS, Pozzilli
  - IRCCS San Raffaele Pisana, Rome
  - Sant'Andrea Hospital, Sapienza University of Rome, Rome
  - University of Turin, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martelletti P, Barbanti P, Grazzi L, Pierangeli G, Rainero I, Geppetti P, Ambrosini A, Sarchielli P, Tassorelli C, Liebler E, de Tommaso M; PRESTO Study Group. Consistent effects of non-invasive vagus nerve stimulation (nVNS) for the acute treatment of migraine: additional findings from the randomized, sham-controlled, double-blind PRESTO trial. J Headache Pain. 2018 Nov 1;19(1):101. doi: 10.1186/s10194-018-0929-0. PMID 30382909
- [Derived] Grazzi L, Tassorelli C, de Tommaso M, Pierangeli G, Martelletti P, Rainero I, Geppetti P, Ambrosini A, Sarchielli P, Liebler E, Barbanti P; PRESTO Study Group. Practical and clinical utility of non-invasive vagus nerve stimulation (nVNS) for the acute treatment of migraine: a post hoc analysis of the randomized, sham-controlled, double-blind PRESTO trial. J Headache Pain. 2018 Oct 19;19(1):98. doi: 10.1186/s10194-018-0928-1. PMID 30340460
- [Derived] Tassorelli C, Grazzi L, de Tommaso M, Pierangeli G, Martelletti P, Rainero I, Dorlas S, Geppetti P, Ambrosini A, Sarchielli P, Liebler E, Barbanti P; PRESTO Study Group. Noninvasive vagus nerve stimulation as acute therapy for migraine: The randomized PRESTO study. Neurology. 2018 Jul 24;91(4):e364-e373. doi: 10.1212/WNL.0000000000005857. Epub 2018 Jun 15. PMID 29907608

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 patients were excluded from the study at the end of the 4-week Run-In/Observational period because they did not continue to meet the study eligibility criteria, were lost to follow-up, or they chose not to continue in the study.
Period: Run-In Period 1
Arm/Group | gammaCore-S | gammaCore-S Sham
Started | 142 | 143
Completed | 122 | 126
Not Completed | 20 | 17
Not completed — Eligibility | 12 | 10
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 4 | 4
Period: Randomized Controlled Period 2
Arm/Group | gammaCore-S | gammaCore-S Sham
Started | 122 | 126
Completed | 117 | 122
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Spontaneous reduction in migraines | 1 | 0
Period: Open Label Period 3
Arm/Group | gammaCore-S | gammaCore-S Sham
Started | 117 | 122
Completed | 117 | 121
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population, n=243
Groups:
- Total: Total of all reporting groups
Arm/Group | gammaCore-S | gammaCore-S Sham | Total
Number analyzed (Participants) | 120 | 123 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (11.00) | 39.6 (11.78) | 39.2 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 91 | 186
  Male | 25 | 32 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 120 | 123 | 243
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 120 | 123 | 243
Age of Onset of Migraine Attacks [Mean (Standard Deviation); unit: years] | 29.42 (11.20) | 28.51 (11.52) | 28.96 (11.35)
Migraine with Aura Diagnosis [Count of Participants; unit: Participants] | 8 | 9 | 17
Number of Migraine Attacks Per Month in Last 6 Months [Mean (Standard Deviation); unit: Attacks per month] | 5.4 (1.51) | 5.4 (1.48) | 5.4 (1.49)
Days Per Month Acute Migraine Medication Taken [Mean (Standard Deviation); unit: Days per month] | 5.6 (1.69) | 5.3 (1.66) | 5.5 (1.68)
Currently Taking Migraine Prevention Medication [Count of Participants; unit: Participants] | 42 | 35 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Response - No Pain
Description: The primary objective is to compare the treatment response for nVNS and Sham therapies at two hours post-treatment, for the first treated migraine attack during study Period 2. Treatment response is defined as no pain at 2 hours post-treatment and no rescue medication use by 2 hours post-treatment.
Time Frame: 2 hours post-treatment
Population: Sensitivity analysis, Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants | 36 | 26

2. Secondary Outcome: Number of Participants With Absence of Nausea/Vomiting, Photophobia, Phonophobia
Description: Presence or absence of nausea/vomiting, photophobia and phonophobia for nVNS and sham therapies for the first treated migraine attack at 120 minutes during study Period 2.
Time Frame: 2 hours post-treatment study - period 2 (each study period was 4 weeks)
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants
  No Nausea at 120 minutes: number analyzed (Participants) | 113 | 116
  No Nausea at 120 minutes | 83 | 86
  No Vomiting at 120 minutes: number analyzed (Participants) | 113 | 115
  No Vomiting at 120 minutes | 110 | 109
  No Photophobia at 120 minutes: number analyzed (Participants) | 113 | 116
  No Photophobia at 120 minutes | 76 | 72
  No Phonophobia at 120 minutes: number analyzed (Participants) | 112 | 116
  No Phonophobia at 120 minutes | 75 | 74

3. Secondary Outcome: Number of Participants With Treatment Response - No Pain or Mild Pain
Description: Response to treatment was assessed by the subjects using the 4 point headache scale, where 0 = No pain, 1 = Mild pain, 2 = Moderate pain and 3 = severe pain.
  Results show count of participants with a response of no pain (score = 0) or mild pain (score = 1) on the 4-point headache pain scale for the nVNS and sham therapies at 2 hours post-treatment and no rescue medication use by 2 hours post-treatment for the first treated migraine attack during study Period 2.
Time Frame: 2 hours post-treatment
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants | 62 | 50

4. Secondary Outcome: Number of Participants With Treatment Response no Pain or Mild Pain at 24 and 48 Hours.
Description: Response to treatment was assessed by the subjects using the 4 point headache scale, where 0 = No pain, 1 = Mild pain, 2 = Moderate pain and 3 = severe pain.
  Results show count of participants with a response of no pain or mild pain on the 4-point headache pain scale at 24, and 48 hours post-treatment (and no rescue medication use) for nVNS and sham therapies for the first treated migraine attack during study Period 2.
Time Frame: 24 and 48 hours post-treatment
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants
  24 Hours | 46 | 37
  48 Hours | 43 | 33

5. Secondary Outcome: Number of Migraine Attacks With Treatment Response 'No Pain' in Study Period 2 All Attacks
Description: Response to treatment was assessed by the subjects using the 4 point headache scale, where 0 = No pain, 1 = Mild pain, 2 = Moderate pain and 3 = severe pain.
  Results show % Treatment response 'No pain' for the nVNS and sham therapies at 30, 60 and 120 minutes calculated for all treated attacks during study Period 2.
Time Frame: 30, 60, 120 minutes; Study Period 2 (each study period was 4 weeks)
Population: Intent to Treat
Measure: Count of Units; unit: Attacks
Units Other Than Participants: Attacks
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Number analyzed (Attacks) | 373 | 347
Attacks
  30 Minutes | 43 | 28
  60 Minutes | 69 | 41
  120 Minutes | 93 | 66

6. Other Pre Specified Outcome: Number of Migraine Attacks With Treatment Response 'No Pain' in Study Period 3
Description: Response to treatment was assessed by the subjects using the 4 point headache scale, where 0 = No pain, 1 = Mild pain, 2 = Moderate pain and 3 = severe pain.
  Number of migraine attacks with treatment response 'no pain' for the nVNS and sham therapies at 30, 60 and 120 minutes calculated for all treated attacks during study Period 3.
Time Frame: 30, 60, 120 minutes; Period 3 (each study period was 4 weeks)
Population: Intent to Treat Period 2 373/347 attacks treated Period 3 286/309 attacks treated
Measure: Count of Units; unit: Attacks
Units Other Than Participants: Attacks
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 117 | 122
Number analyzed (Attacks) | 286 | 309
Attacks
  30 Minutes | 35 | 41
  60 Minutes | 47 | 61
  120 Minutes | 63 | 83

7. Other Pre Specified Outcome: Number of Migraine Attacks With Treatment Response no Pain or Mild Pain
Description: Response to treatment was assessed by the subjects using the 4 point headache scale, where 0 = No pain, 1 = Mild pain, 2 = Moderate pain and 3 = severe pain.
  Number of migraine attacks with treatment response 'no pain' or 'mild pain' on the 4-point headache pain scale for the nVNS and sham therapies at 30, 60 and 120 minutes calculated for all treated attacks during study Periods 2 and 3 (separately)
Time Frame: 30, 60, 120 minutes; Study Periods 2 and 3 (each study period was 4 weeks)
Population: Intent to Treat Period 2 373/347 attacks treated Period 3 286/309 attacks treated
Measure: Count of Units; unit: Attacks
Units Other Than Participants: Attacks
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Number analyzed (Attacks) | 373 | 347
Attacks
  Period 2 30 Minutes | 149 | 123
  Period 2 60 Minutes | 160 | 130
  Period 2 120 Minutes | 165 | 136
  Period 3 30 Minutes: number analyzed (Participants) | 117 | 122
  Period 3 30 Minutes: number analyzed (Attacks) | 286 | 309
  Period 3 30 Minutes | 105 | 122
  Period 3 60 Minutes: number analyzed (Participants) | 117 | 122
  Period 3 60 Minutes: number analyzed (Attacks) | 286 | 309
  Period 3 60 Minutes | 117 | 140
  Period 3 120 Minutes: number analyzed (Participants) | 117 | 122
  Period 3 120 Minutes: number analyzed (Attacks) | 286 | 309
  Period 3 120 Minutes | 124 | 147

8. Other Pre Specified Outcome: Number of Migraine Attacks With Absence of Nausea, Vomiting, Photophobia and Phonophobia
Description: Number of Attacks with Absence of Nausea, Vomiting, Photophobia and Phonophobia at 120 minutes for nVNS and sham therapies calculated for all treated attacks during study Periods 2 and 3 (separately).
Time Frame: Study Periods 2 and 3 (each study period was 4 weeks)
Population: Intent to Treat population Period 2 373/347 attacks treated Period 3 286/309 attacks treated
Measure: Count of Units; unit: Attacks
Units Other Than Participants: Attacks
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Number analyzed (Attacks) | 373 | 347
Attacks
  No Nausea Period 2 | 253 | 228
  No Vomiting Period 2 | 342 | 312
  No Photophobia Period 2 | 233 | 202
  No Phonophobia Period 2 | 223 | 203
  No Nausea Period 3: number analyzed (Participants) | 117 | 122
  No Nausea Period 3: number analyzed (Attacks) | 286 | 309
  No Nausea Period 3 | 195 | 226
  No Vomiting Period 3: number analyzed (Participants) | 117 | 122
  No Vomiting Period 3: number analyzed (Attacks) | 286 | 309
  No Vomiting Period 3 | 268 | 288
  No Photophobia Period 3: number analyzed (Participants) | 117 | 122
  No Photophobia Period 3: number analyzed (Attacks) | 286 | 309
  No Photophobia Period 3 | 158 | 195
  No Phonophobia Period 3: number analyzed (Participants) | 117 | 122
  No Phonophobia Period 3: number analyzed (Attacks) | 286 | 309
  No Phonophobia Period 3 | 154 | 203

9. Other Pre Specified Outcome: Number of Attacks With Sustained Treatment Response
Description: Number of migraine attacks with sustained treatment response (mild or no pain at 24 and 48 hours post-treatment) for nVNS and sham therapies calculated for all treated attacks during study Periods 2 and 3 (separately).
Time Frame: 24 and 48 hours; Study Periods 2 and 3 (each study period was 4 weeks)
Population: Intent to treat Period 2 373/347 attacks treated Period 3 286/309 attacks treated
Measure: Count of Units; unit: Attacks
Units Other Than Participants: Attacks
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Number analyzed (Attacks) | 373 | 347
Attacks
  24 Hours, Period 2 | 132 | 103
  48 Hours, Period 2 | 121 | 95
  24 Hours, Period 3: number analyzed (Participants) | 117 | 122
  24 Hours, Period 3: number analyzed (Attacks) | 286 | 309
  24 Hours, Period 3 | 100 | 117
  48 Hours, Period 3: number analyzed (Participants) | 117 | 122
  48 Hours, Period 3: number analyzed (Attacks) | 286 | 309
  48 Hours, Period 3 | 96 | 111

10. Other Pre Specified Outcome: Number of Subjects With Consistency of Response
Description: Consistency of response, defined as the number of subjects who achieve no pain or mild pain in 50% or greater of their attacks, in subjects treating at least two attacks, for nVNS and sham therapies for all treated attacks during study Periods 2 and 3 (separately).
Time Frame: Study Periods 2 and 3 (each study period was 4 weeks)
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
participants
  Period 2 | 57 | 46
  Period 3: number analyzed (Participants) | 117 | 122
  Period 3 | 44 | 44

11. Other Pre Specified Outcome: Quality of Life Measured by EuroQol-5D-5L (EQ-5D-5L)
Description: Treatment effect on quality of life: EQ-5D-5L is assessed at end of the run-in period and at the end of each 4-week period for nVNS and sham therapies.
  EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1 = no problems, 2 = slight problems, 3= moderate problems, 4 = severe problems and 5 = extreme problems. Subjects indicate health state by ticking choosing appropriate statement in each dimension. The 5 dimensions scores are combined into a score, where a lower score indicates less problems.
  Scores across all 5 dimensions are averaged resulting in a total theoretical score of 1 to 5 with lower scores indicating less problems
Time Frame: End of each study period (each study period was 4 weeks)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 142 | 143
Score
  EQ5D5L - Visit 1 Start of run-in period | 0.885 (0.1028) | 0.912 (0.0969)
  EQ5D5L - Visit 3 End of run-in period: number analyzed (Participants) | 122 | 126
  EQ5D5L - Visit 3 End of run-in period | 0.896 (0.0903) | 0.917 (0.0980)
  EQ5D5L -Visit 5 End of randomised period: number analyzed (Participants) | 117 | 122
  EQ5D5L -Visit 5 End of randomised period | 0.911 (0.0980) | 0.926 (0.0951)
  EQ5D5L - Visit 7 End of open label period: number analyzed (Participants) | 117 | 121
  EQ5D5L - Visit 7 End of open label period | 0.923 (0.0924) | 0.931 (0.0910)

12. Other Pre Specified Outcome: Bang Blinding Index Scores
Description: After the first treated attack and at the end of the double blind period (period 2) subjects were asked to guess if they were had received 'gammaCore-S', ''sham' or 'do not know'. Bang blinding index estimated are presented for the gammaCore-S and sham.
  Bang Blinding Index shows the success of blinding. The blinding index proposed is scaled to an interval of -1 to 1, 1 being complete lack of blinding, 0 being consistent with perfect blinding and -1 indicating opposite guessing which may be related to unblinding.
  A score of one means they guess correctly, -1 incorrectly. If the bang index includes 0 it indicates that the guesses were consistent for the sham and active and the study was appropriately blinded
Time Frame: Study Period 2 (4 weeks)
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: Bang Blinding Index Score
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Bang Blinding Index Score
  First Treated Attack | 0.07 [-0.037 to 0.173] | 0.00 [-0.106 to 0.106]
  End of Period 2 | -0.03 [-0.143 to 0.075] | 0.23 [0.125 to 0.334]

13. Other Pre Specified Outcome: Subject Satisfaction
Description: Subject satisfaction with the study devices Subjects were asked to rate their satisfaction with the device from the following options: Extremely satisfied, Very satisfied, Satisfied, A little satisfied or Not at all satisfied
Time Frame: End of Study Periods 2 and 3 (each study period was 4 weeks long)
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants
  Visit 5 Extremely Satisfied | 7 | 8
  Visit 5 Very Satisfied | 18 | 12
  Visit 5 Satisfied | 27 | 22
  Visit 5 A Little Satisfied | 33 | 36
  Visit 5 Not at All Satisfied | 33 | 44
  Visit 7 Extremely Satisfied | 10 | 12
  Visit 7 Very Satisfied | 19 | 18
  Visit 7 Satisfied | 23 | 34
  Visit 7 A Little Satisfied | 32 | 26
  Visit 7 Not at All Satisfied | 31 | 28

14. Other Pre Specified Outcome: Mean Change in Pain Score From Baseline to 120 Minutes
Description: Subjects rated pain at onset of migraine attack (baseline) and at 120 minutes using a 4 point headache pain scale where 0 = no pain, 1 = mild pain, 3 = moderate pain and 4 = severe pain. A lower score indicates less pain. Mean change in pain score from baseline to 120 minutes for all attacks in study period 2
Time Frame: 120 minutes, Study Period 2 (each study period was 4 weeks long)
Population: Intent to Treat
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
score on a scale | -0.4954 [-0.6509 to -0.3399] | -0.2769 [-0.4392 to -0.1146]

15. Other Pre Specified Outcome: Ease of Use
Description: Ease of use of the study devices - Subjects were asked to rate the ease of use of the device from the following options: Very easy, somewhat easy, difficult, very difficult.
Time Frame: End of Study Periods 2 and 3 (each study period was 4 weeks long)
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 120 | 123
Participants
  Visit 5 Very Easy: number analyzed (Participants) | 118 | 122
  Visit 5 Very Easy | 90 | 97
  Visit 5 Easy: number analyzed (Participants) | 118 | 122
  Visit 5 Easy | 23 | 20
  Visit 5 Difficult: number analyzed (Participants) | 118 | 122
  Visit 5 Difficult | 5 | 4
  Visit 5 Very Difficult: number analyzed (Participants) | 118 | 122
  Visit 5 Very Difficult | 0 | 1
  Visit 7 Very Easy: number analyzed (Participants) | 115 | 118
  Visit 7 Very Easy | 92 | 98
  Visit 7 Easy: number analyzed (Participants) | 115 | 118
  Visit 7 Easy | 18 | 17
  Visit 7 Difficult: number analyzed (Participants) | 115 | 118
  Visit 7 Difficult | 5 | 3
  Visit 7 Very Difficult: number analyzed (Participants) | 115 | 118
  Visit 7 Very Difficult | 0 | 0

16. Other Pre Specified Outcome: Quality of Life Measured by Headache Impact Test (HIT-6)
Description: The HIT-6 measures impact of headaches on ability to function at work, at home and in social situations. Subjects answer 6 questions about ability to function and normal daily life and for each question they rate the impact of their headaches as 'never' (6 points) or 'rarely' (9 points) or 'sometimes' (10 points) or 'very often' (11 points) or 'always' (13 points). Minimum score = 36, maximum score = 78.
  Higher score is worse and lower score is better quality of life
Time Frame: End of each study period (each study period was 4 weeks)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | gammaCore-S | gammaCore-S Sham
Number analyzed (Participants) | 142 | 143
Score
  HIT6 - Visit 1 Start of run-in period | 63.250 (5.0581) | 63.179 (5.2977)
  HIT6 - Visit 3 End of run-in period: number analyzed (Participants) | 122 | 126
  HIT6 - Visit 3 End of run-in period | 63.275 (5.4618) | 61.894 (5.5704)
  HIT6 - Visit 5 End of randomised period: number analyzed (Participants) | 117 | 122
  HIT6 - Visit 5 End of randomised period | 61.897 (5.5900) | 60.959 (5.6604)
  HIT6 - Visit 7 End of open label period: number analyzed (Participants) | 117 | 121
  HIT6 - Visit 7 End of open label period | 61.128 (5.5871) | 60.750 (5.7149)

ADVERSE EVENTS:
Time Frame: 12 weeks - Period 1 (4 weeks), Period 2 (4 weeks) and Period 3 (4 weeks)
Arm/Group | gammaCore-S | gammaCore-S Sham
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/126
Other Adverse Events (participants affected / at risk) | 22/122 | 23/126
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore-S (N=122) | gammaCore-S Sham (N=126)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (2) | 0 (0)
Application site discomfort (General disorders) | 3 (3) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 3 (5)
Application site hyperaesthesia (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 0 (0) | 3 (4)
Application site paraesthesia (General disorders) | 0 (0) | 1 (1)
Application site rash (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Blood pressure (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Status migrainosus (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Varicocele repair (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less